CLINICAL TRIAL: NCT04036643
Title: Contribution of [18F] -FDG-PET / MRI in the Detection of the Absence of Complete Response After Neo-adjuvant Radiotherapy for Cancers of the Middle and Low Rectum for a Treatment Procedure With Rectal Savings
Brief Title: Rectal Cancer Response Hybrid Imaging Assessement
Acronym: RECARHIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P170939J
Record Dates: First submitted 2019-07-01; First posted 2019-07-30 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Rectal Cancer
Keywords: Rectal neoplasm; Imaging TEP/MRI; response assessement
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: All patient with rectal cancer treated by neoadjuvant chemo radiation therapy with clinical complete response
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with rectal cancer (Experimental): Patient with rectal cancer treated by neoadjuvant chemo-radiation therapy with clinical complete response
  Interventions: Radiation: PET-MRI

INTERVENTIONS:
Radiation: PET-MRI — Hybrid PET / MRI machine for simultaneous acquisition of functional and molecular information of different natures coupled with the high anatomical resolution of MRI.

SUMMARY:
Rectal cancer represents 14,000 new cases a year in France. At diagnosis, 70% of patients have a locally advanced tumors T3-T4 and / or N + evaluated mainly by rectal MRI. These patients will benefit from a neo-adjuvant treatment by radio-chemotherapy. The complete histologic response rate (ypT0N0) after this neo-adjuvant treatment ranged from 15 to 27% and improved recurrence-free survival, remotely relapse-free survival, overall survival, and decreased local recurrence rate. In the case of full response diagnosis after neoadjuvant chemoradiotherapy 3 theoretical solutions exist:

1. Total excision of the rectum and mesorectum (TME) This is the classic attitude with a low risk of local recurrence (5%) but functional complications occur in 25 to 60% of cases
2. A simple monitoring ("Watch and Wait") by MRI, biopsy, rectoscopy ... This strategy was initially proposed to elderly patients considered inoperable but it has also been proposed in younger patients, operable, with a view to decreasing morbidity and sequelae. This attitude poses a likely overall risk of local recidivism. However, this higher risk of recurrence may be the result of imperfect identification of ypT0N0 patients.
3. Local excision of the post-radiation scar also called closure lumpectomy with pathological analysis and possible secondary TME if no complete response. This last attitude has the advantage of allowing an anatomopathological verification of the treated lesion and to complete the treatment if necessary. In the case of ypT0 the local recurrence rate is low and in this case it is possible to consider rectal savings.

The choice of the last two attitudes is therefore based on the correct identification of patients in complete response. The performance of the diagnosis of no complete response after radiochemotherapy is therefore fundamental and is the subject of this project wich consist of comparing he diagnostic performance for the identification of a complete lack of response [18F] -FDG-PET / MRI ypT0N0 to that of the classic attitude (MRI) 6 to 9 weeks after the end of a neoadjuvant chemoradiotherapy treatment of low and mid-rectal cancers in patients in whom clinical and endoscopic examination favor a complete response.

DETAILED DESCRIPTION:
The MRI examination to evaluate the response to routine Radio-Chemotherapy Neoadjuvant (RCT) will be replaced by an MRI-PET scan in all patients included. Firstly, only the MRI portion of the examination will be interpreted (sequences identical to that performed in conventional MRI), without the PET part of the examination. An evaluation of the answer will be done. The results of the MRI will be transmitted to the surgeon in accordance with the conventional attitude of treatment of rectal cancer treated with RCT.

In a second step the complete examination associating the merged MRI and PET sequences will be reinterpreted. A new evaluation of the response will be done. The results of the MRI and PET MRI will be read without the gold standard, which will be available after the intervention. The results of this second analysis will not be transmitted to the Multidisciplinary Concertation Meeting and will not influence the management. The patients will then be operated. The histological stage ypTN will be established on the operative specimen.

Thus all patients will have the 2 tests under study (MRI and [18F] -FDG-PET / MRI, as well as the gold standard (pathological analysis) .These results will meet the main objective evaluation of the diagnostic performances by comparing them with the results of the gold standard (anatomopathological analysis of the operative specimen)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age ≥18 years
* Patients with a rectal cancer and who had neo-adjuvant treatment by radio-chemotherapy
* Patients for whom the clinical and endoscopic examination realised 6 at 9 weeks after the end o the RCT is in favour of a complete response (normal digital rectal exam, endoscopic complete disappearance of the lesion or the presence of scar and whitish plane of less than 2 cm)
* Patients who have signed a consent formulary after a loyal and fair information
* Patients affiliated to a social security scheme (beneficiary or legal) outside AME

Exclusion Criteria:

* Patients with a contraindication to MRI: pacemaker, defibrillator, intraocular metallic foreign body, ferromagnetic implant, claustrophobia
* Patient with a contraindication to PET: non controlled diabet glycemia > 200 mh/dL, pregnancy
* Hypersensibility to 18-FDG or others contrast products
* Patients who would require abdominoperineal amputation
* Patients with many comorbidities contraindicating MTCT because these patients do not match the target population (in addition they currently represent the rare indications of closure lumpectomy)
* Patients under guardianship or reinforced curators or deprived of liberty.
* Pregnant or childbearing women without effective contraception (a plasma βHCG test will be performed in this case the day before PET / MRI)
* Participation in another interventional research without the agreement of the physician following the patient for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-11-27 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Tumor response assessed by modified the Ryan tumor regression grading system obtained by quantification of the residual cancer cells compared to fibrosis on the surgical specimen | Up to 3 months
  After surgery the tumor response will be graded TRG 1 (no residual cancer cells), 2 (residual cancer outgrown by fibrosis) or 3 (fibrosis outgrown by cancer cells). MRI and [18F] -FDG-PET / MRI results (residual tumor or no residual tumor) will be compared to TRG results and Sensitivity and specificity of MRI and [18F] -FDG-PET / MRI for TRG1 will be calculated

SECONDARY OUTCOMES:
Calculation of the Net Reclassification Index (NRI) by comparing the sensitivity of [18F] -FDG-PET / MRI and the sensitivity of MRI alone for TRG1 | Up to 3 months
  Number of patient correctly reclassified with [18F] -FDG-PET as having a complete response (no residual tumor visible) divided by the number of patient correctly classified with [18F] -FDG-PET as having a complete response (no residual tumor visible)

CONTACTS AND LOCATIONS:
Overall Officials: LUCIDARME Olivier, PU-PH, Principal Investigator — AP-HP Groupe Hospitalier Pitié Salpêtrière - Radiology Department
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France